CLINICAL TRIAL: NCT06075771
Title: Dopaminergic Therapy for Inflammation-Related Anhedonia in Depression - 2
Brief Title: Dopaminergic Therapy for Anhedonia - 2
Acronym: DTA-2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jennifer Felger, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00006669; R33MH121625-02 (NIH)
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Anhedonia; Depression
Keywords: Anhedonia; Depression
MeSH Terms: conditions — Anhedonia; Depression | interventions — carbidopa, levodopa drug combination; Levodopa

STUDY DESIGN:
Intervention Model Description: 2:1 randomization to L-DOPA versus placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carbidopa Levodopa Group (Experimental): Patients randomized to the Carbidopa Levodopa Group will receive one tablet per day of L-DOPA (150 mg levodopa administered with 37.5 mg carbidopa) for 4 weeks.
  Patients that respond after the initial 4 weeks will continue on the same dose for an additional 4 weeks to determine whether clinical response at the 150 mg dose is sustained over time compared to placebo.
  Patients that do not exhibit a clinical response (50% reduction in HAM-D scores from baseline) after 4-weeks on the 150 mg dose will escalate to 450 mg L-DOPA (three tablets per day of 150 mg levodopa administered with 37.5 mg carbidopa) and studied over an additional 4 weeks (8 weeks total in the study).
  Interventions: Drug: Carbidopa Levodopa
- Placebo Group (Placebo Comparator): Participants will receive placebo tablet. Placebo-treated non-responders at 4 weeks will remain on placebo but with the same instructions to increase daily pill intake.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carbidopa Levodopa — Patients will receive between one and three tablets per day of 150 mg L-DOPA (administered with 37.5 mg carbidopa) to achieve doses ranging from 150 to 450 mg/day.
  Other Names: Sinemet, L-DOPA
  Arms: Carbidopa Levodopa Group
Drug: Placebo — A placebo is a sugar pill that has no therapeutic effect and will be administered orally. Participants will receive between one and three placebo tablets per day matching the Carbidopa Levodopa tablet.
  Other Names: Placebo tablet
  Arms: Placebo Group

SUMMARY:
The purpose of this 8-week, double-blind, placebo-controlled, study is to explore new treatment options for people with depression who have high inflammation and anhedonia. Seventy male and female participants with depression, between 25-55 years of age, with higher levels of inflammation and anhedonia will be randomized to receive L-DOPA or matched placebo over 8 weeks. Participants will complete lab tests, medical and psychiatric assessments, motivation and motor tasks, and MRI scans as part of the study. The total length of participation is approximately 10 to 12 weeks.

DETAILED DESCRIPTION:
Depression is a widespread disorder (lifetime prevalence >20%). Current antidepressant medications are effective for many patients; however, more than 30% fail to respond. Of the patients that do respond to treatment, some continue to suffer with primary symptoms of depression like an inability to experience pleasure, called anhedonia. In this regard, one biological pathway that may contribute to symptoms of depression and particularly anhedonia is inflammation.

The purpose of this 8-week, double-blind, placebo-controlled, study is to explore new treatment options for people with depression who have high inflammation and anhedonia. Despite evidence of low dopamine function in patients with depression, the ability of existing dopaminergic therapies, like L-DOPA, to affect brain circuits in depression has yet to be explored. This study will help determine whether an FDA-approved medication, Sinemet (L-DOPA), might be used in the future to treat sub-groups of depressed individuals.

Seventy male and female participants with depression, between 25-55 years of age, with higher levels of inflammation and anhedonia will be randomized to receive L-DOPA or matched placebo over 8 weeks. Participants will complete lab tests, medical and psychiatric assessments, motivation and motor tasks, and MRI scans as part of the study. The total length of participation is approximately 10 to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* a. willing and able to give written informed consent
* b. men or women, 25-55 years of age
* c. a primary diagnosis of Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), current, as diagnosed by the Structured Clinical Interview for DSM-5
* d. score of >10 on the Patient Health Questionnaire-9 (PHQ-9) or HAM-D score ≥18
* e. off all antidepressant or other psychotropic therapy (e.g. mood stabilizers, antipsychotics, anxiolytics, and sedative hypnotics) for at least 4 weeks prior to baseline visit (8 weeks for fluoxetine)
* f. c-reactive protein (CRP) ≥2 mg/L
* g. PHQ-9 anhedonia score ≥2

Exclusion Criteria:

* a. history or evidence (clinical or laboratory) of an autoimmune disorder
* b. history or evidence (clinical or laboratory) of hepatitis B or C infection or human immunodeficiency virus infection
* c. history of any type of cancer requiring treatment with more than minor surgery
* d. unstable cardiovascular, endocrinologic, hematologic, hepatic, renal, or neurologic disease (as determined by physical examination, EKG and laboratory testing)
* e. history of any (non-mood-related) psychotic disorder; active psychotic symptoms of any type; history or current bipolar disorder; history or current gambling disorder; substance abuse/dependence within 6 months of study entry (as determined by standardized clinician interview)
* f. active suicidal plan as determined by a score >3 on item #3 on the HAM-D
* g. an active eating disorder (except for patients with binge eating disorder in whom binging is clearly associated with worsening of mood symptoms)
* h. a history of a cognitive disorder or traumatic head injury involving loss of consciousness
* i. pregnancy or lactation
* j. use of gender affirming hormone therapy
* k. chronic use of non-steroidal anti-inflammatory agents (NSAIDS) (excluding 81mg of aspirin), glucocorticoid containing medications or statins
* l. use of NSAIDS, glucocorticoids, or statins at any time during the study
* m. urine toxicology screen is positive for drugs of abuse, n. any contraindication for MRI scanning
* o. intolerance, sensitivity or contraindication to carbidopa-levodopa (including history of narrow-angle glaucoma, melanoma, gastric and/or duodenal ulcers, bleeding disorders, or frequent migraines)

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptom severity measured by Hamilton Depression Rating Scale (HAM-D) | Baseline, weeks 1-4 post-intervention, weeks 5-8 post-intervention
  The HAM-D-17 is a 17-item, clinician administered scale, that rates severity of depression. Each item is rated on a scale 0-4 with higher scores indicating greater pathology.

SECONDARY OUTCOMES:
Change in corticostriatal functional connectivity (FC) in reward circuits | Baseline, week 4 post-intervention, week 8 post-intervention
  Patients will undergo resting-state and task-based functional magnetic resonance imaging (fMRI) to calculate functional connectivity (FC) between the ventral striatum (VS) and ventromedial prefrontal cortex (vmPFC). FC is measured as continuous Z scores reflecting the correlation of activity between the brain regions. Higher FC Z scores reflect stronger connectivity.
Change in objective motivation assessed by Effort-Expenditure for Rewards Task (EEfRT) | Baseline, week 4 post-intervention, week 8 post-intervention
  The EEfRT is a widely used, multi-trial task in which participants are given an opportunity on each trial to choose between two different task difficulty levels in order to obtain monetary rewards. EEfRT will be used as an objective measure of motivation, and will be administered following MRI scans during the study. The EEfRT is reported as the percent of high effort trials selected. A higher percentage reflects higher motivation for effort expenditure.
Change in Inventory of Depressive Symptomatology- Self-Report (IDS-SR) | Baseline, weeks 1-4 post-intervention, weeks 5-8 post-intervention
  Anhedonia will be assessed from a subscale of the IDS-SR. Scores on this 3-question scale range from 0-9 with higher scores reflecting greater anhedonia.
Change in Snaith-Hamilton Pleasure Scale-Clinician (SHAPS-C) | Baseline, weeks 1-4 post-intervention, weeks 5-8 post-intervention
  The SHAPS-C is a clinician administered tool to assess symptoms of anhedonia. The SHAPS-C uses14 questions each rated on a Likert scale of 1-4, with higher scores reflecting greater pathology.
Change in Motivation and Pleasure-Self-Report (MAP-SR) | Baseline, weeks 1-4 post-intervention, weeks 5-8 post-intervention
  The MAP-SR will be used to capture self-reported aspects of anhedonia and reduced motivation. The scale uses 18 questions each rated on a Likert scale of 0-4, with higher scores reflecting greater pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Felger, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Only the data - raw and analyzed, or both, depending on the items. Statistical plans an additional information may be shared within the data base but it is not required as the data will be linked to the publications.
Supporting Information: SAP
Time Frame: After publication, within one year of the end of the project.
Access Criteria: Must be NIH investigators and they have to submit an application, including analysis plan, in order to be granted access.